CLINICAL TRIAL: NCT07368387
Title: The Effect of QR Code-Based Preoperative Education on Anxiety, Postpartum Pain, and Comfort in Women Undergoing Cesarean Birth
Brief Title: QR Code-Based Preoperative Education for Cesarean Birth: Anxiety, Pain, and Comfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Reyhan Aydin Doğan, ASSOCIATE PROFESSOR, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/1494
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Preoperative Anxiety; Postpartum Pain; Maternal Comfort; Cesarean Birth
Keywords: Cesarean Birth; Preoperative Education; QR Code-Based Education; Maternal Anxiety; Postpartum Pain; Maternal Comfort; Digital Health Education; Randomized Controlled Trial; Prenatal Education

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: an intervention group receiving QR code-based preoperative education and a control group receiving routine preoperative care. Each participant will be exposed to only one study condition throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QR Code-Based Preoperative Education (Experimental): Participants in this arm will receive structured preoperative education delivered through QR code-based digital materials prior to elective cesarean birth. The educational content will include information about the cesarean procedure, perioperative expectations, postoperative pain management, and comfort-enhancing strategies.
  Interventions: Behavioral: QR Code-Based Preoperative Education
- Control (No Intervention): Participants in this arm will receive routine preoperative care and standard information provided by the hospital without access to the QR code-based educational materials.

INTERVENTIONS:
Behavioral: QR Code-Based Preoperative Education — Educational intervention delivered via QR code-based digital materials providing preoperative information on cesarean birth, postoperative pain management, and comfort strategies.
  Arms: QR Code-Based Preoperative Education

SUMMARY:
This study aims to evaluate the effect of QR code-based preoperative education on anxiety, postpartum pain, and comfort levels in women undergoing cesarean birth. Cesarean delivery is a common surgical procedure, and insufficient preoperative information may increase anxiety and negatively affect postoperative recovery and comfort.

In this randomized controlled study, eligible pregnant women scheduled for elective cesarean birth will be assigned to either an intervention group or a control group. Women in the intervention group will receive preoperative education delivered through QR code-based digital materials, including information about the cesarean procedure, postoperative pain management, and comfort-enhancing strategies. The control group will receive routine care provided by the hospital.

Anxiety levels will be assessed preoperatively, while postpartum pain and comfort levels will be evaluated after delivery using validated measurement tools. The findings of this study are expected to contribute to the development of accessible and effective educational interventions to improve maternal well-being and postoperative outcomes in cesarean birth.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to examine the effects of QR code-based preoperative education on anxiety, postpartum pain, and comfort among women undergoing elective cesarean birth. The study will be conducted in a hospital setting and will include pregnant women who meet the predefined inclusion criteria and provide informed consent.

Participants will be randomly allocated into two groups: an intervention group and a control group. Randomization will be performed using a predetermined allocation method to ensure comparability between groups. Women assigned to the intervention group will receive structured preoperative education delivered through QR code-based digital materials. These materials will include information on the cesarean birth process, perioperative expectations, postoperative pain management, and strategies to enhance physical and psychological comfort. Participants will be able to access the educational content using their personal mobile devices prior to surgery. The control group will receive routine preoperative care and standard information provided by the hospital.

Data collection will be carried out at multiple time points. Preoperative anxiety levels will be assessed prior to the cesarean procedure. Postpartum pain and comfort levels will be evaluated after delivery during the postoperative period. Validated measurement instruments will be used to collect outcome data. Sociodemographic and obstetric characteristics will also be recorded to describe the study population and to control for potential confounding variables.

The primary outcomes of the study are changes in preoperative anxiety and postoperative pain and comfort levels. The study does not involve the use of any pharmacological agents or medical devices and poses minimal risk to participants. The results are expected to provide evidence on the effectiveness of digital, easily accessible educational interventions in improving maternal outcomes in cesarean birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older
* Scheduled for elective (planned) cesarean birth
* Able to read and understand Turkish and complete study questionnaires
* Able to provide written informed consent
* Has access to a smartphone and is able to use a QR code to view the educational materials (intervention arm)

Exclusion Criteria:

* Emergency cesarean birth or unplanned change to emergency surgery
* Presence of high-risk pregnancy or serious obstetric/medical complications requiring intensive management (e.g., severe preeclampsia/eclampsia, major hemorrhage risk, unstable systemic disease)
* Known psychiatric disorder or current use of medications that may substantially affect anxiety assessment (as judged by the clinical team)
* Communication barriers that prevent participation (e.g., severe visual/hearing impairment, cognitive impairment) or inability to complete questionnaires
* No smartphone access or inability/unwillingness to use QR code materials (for intervention delivery)
* Refusal to participate or withdrawal of consent at any time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Postpartum Pain Level | Postpartum period following cesarean birth
  Postpartum pain levels will be evaluated to determine the effect of QR code-based preoperative education on pain experienced after cesarean birth. Pain will be assessed using a validated pain assessment tool.
Preoperative Anxiety Level | Preoperatively, prior to cesarean birth
  Preoperative anxiety will be assessed to evaluate the effect of QR code-based preoperative education on anxiety levels in women undergoing elective cesarean birth. Anxiety will be measured using a validated self-report instrument.

SECONDARY OUTCOMES:
Maternal Comfort Level | Postpartum period following cesarean birth
  Maternal comfort will be assessed to examine the effect of QR code-based preoperative education on physical and psychological comfort after cesarean birth. Comfort levels will be measured using a validated comfort assessment scale.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive personal and health-related information collected within a single-center, thesis-based research project. Data confidentiality and participant privacy will be strictly protected in accordance with ethical approval and institutional policies. De-identified, aggregate results will be reported in publications.

REFERENCES:
- [Background] Togac HK, Yilmaz E. Effects of preoperative individualized audiovisual education on anxiety and comfort in patients undergoing laparoscopic cholecystectomy: randomised controlled study. Patient Educ Couns. 2021 Mar;104(3):603-610. doi: 10.1016/j.pec.2020.08.026. Epub 2020 Aug 28. PMID 32933794
- [Background] Mostafayi M, Imani B, Zandi S, Jongi F. The effect of familiarization with preoperative care on anxiety and vital signs in the patient's cesarean section: A randomized controlled trial. Eur J Midwifery. 2021 Jun 25;5:21. doi: 10.18332/ejm/137366. eCollection 2021. PMID 34222839
- [Background] Abuzaid M, Alshahrani MS, Ahmed AM, Moafa MN, Alomar O, O'Mahony A, Abu-Zaid A. Effectiveness of preoperative multimedia educational sessions on the levels of anxiety and satisfaction among women undergoing cesarean: a systematic review and meta-analysis. Women Health. 2024 May-Jun;64(5):416-426. doi: 10.1080/03630242.2024.2349560. Epub 2024 May 5. PMID 38706246